CLINICAL TRIAL: NCT04496180
Title: Standard Wound Dressing Versus Prophylactic Negative-pressure Wound Therapy After Emergency Laparotomy: a Randomized Controlled Trial
Brief Title: Prevena to Prevent Surgical Site Infection After Emergency Abdominal Laparotomy
Acronym: CiPNT/SSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Geneva (Other)
Collaborators: Meyer Jeremy. PhD. Co-investigator. University Hospital, Geneva. (Unknown); Peloso Andrea. PhD. Co-investigator. University Hospital, Geneva. (Unknown); Ris Frederic. P.D. Clinical Professor. University Hospital, Geneva. (Unknown); Toso Christian. PhD. Head of visceral surgery. University Hospital, Geneva. (Unknown); Buchs C. Nicolas. P.D. Director of the project. University Hospital, Geneva. (Unknown)
Responsible Party: Principal Investigator, Abbassi Ziad, Principal investigator, M.D., University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UNGeneva
Record Dates: First submitted 2020-07-16; First posted 2020-08-03 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Surgical Site Infection; Length of Stay; Seroma; Hematoma
Keywords: pNPWT; PREVENA; SSI; morbidity; dehiscence
MeSH Terms: conditions — Surgical Wound Infection; Seroma; Hematoma

STUDY DESIGN:
Intervention Model Description: * Study Type: Interventional (Clinical Trial)
  * Estimated Enrollment: 334
  * Allocation: Randomized control trial
  * Intervention Model: Parallel Assignment
  * Intervention Model Description: 2 separate treatment arms
  * Primary Purpose: Prevention
  * Official Title: Standard wound dressing versus prophylactic negative-pressure wound therapy after emergency laparotomy
  * Estimated Study Start Date: 09.2020
  * Estimated Primary Completion Date:09.2021
  * Estimated Study Completion Date: 09.2025
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PREVENA (CiPNT) (Experimental): Target population is every patient undergoing a laparotomic procedure and responding to inclusion criteria marked in paragraph 3.8 (see forward) A member of the medical surgery team should apply all parts just after the surgical procedure.
  A medical member (nurse specialist in wound care) of the surgical team removes the dressing. All other manipulations of the therapy unit, the connector and the cartridge can be carried out by any nurse practitioner in hospital or extra hospital environment but must warn the investigators.
  The aspiration will be stopped 24 hours before and the dressing is removed by a nurse at home or in the hospital.
  The specialized nurse who will take a photo and assess the condition of the wound in the treatment room.
  One of the investigators, non-operators, who will also assess the condition of the wound by photo.
  Interventions: Device: Closed incision negative pressure therapy versus standard dressing after emergency abdominal laparotomies
- Simple dressing (Active Comparator): Simple dressing; standard, waterproof dressing applied to wound
  Interventions: Device: Closed incision negative pressure therapy versus standard dressing after emergency abdominal laparotomies

INTERVENTIONS:
Device: Closed incision negative pressure therapy versus standard dressing after emergency abdominal laparotomies — Target population is every patient undergoing a laparotomic procedure and responding to inclusion criteria marked in paragraph 3.8 (see forward) A member of the medical surgery team should apply the PREVENA just after the surgical procedure.
  A medical member (nurse specialist in wound care) of the surgical team removes the dressing. All other manipulations of the therapy unit, the connector and the cartridge can be carried out by any nurse practitioner in hospital or extra hospital environment but must warn the investigators.
  The aspiration will be stopped 24 hours before and the dressing is removed by a nurse at home or in the hospital.
  The specialized nurse who will take a photo and assess the condition of the wound in the treatment room.
  One of the investigators, non-operators, who will also assess the condition of the wound by photo.
  Other Names: PREVENA

SUMMARY:
Post-operative wound complications in abdominal surgery have a major impact on patient outcomes and the real impact of Closed incision negative pressure therapy (CINVt) is not clear in the literature moreover concerning its potential economic benefits The hypothesis of this study is that CINPt has the potential to reduce Surgical Site Infections.

Secondly the investigators aim to study the economic impact of CINPt used after abdominal emergency laparotomies.

DETAILED DESCRIPTION:
Emergency laparotomies lead to increased morbidity and mortality rates. In this scenario the most frequent wound occurrences are represented by wound infections, skin dehiscence or parietal hernias.

Despite standard surgical aseptically technique and perioperative prevention management of infections (e.g. antibiotics), wound complications after emergency laparotomies are still an important unmet challenge.

Moreover, all these complications increase the cost of care requiring new managements.

CINPt has been longly used to favour the successful healing of a plethora of open wounds.

In particular CINPt is based on the application of local negative pressure to the wound surface. In case of open abdomens, the procedure is performed by applying a sterile abdominal dressing, which consists of a fenestrated soft plastic non-adherent layer with enclosed central foam, which is placed on the surface of the viscera. Then, two layers of porous sponge dressings are applied over the plastic layer. Finally, a transparent adhesive is placed over the foam and the wound to seal the abdominal cavity. The entire system is then connected, by suction tubes, to a device which ubiquitously applies negative pressure (cyclically or continuously) on the surface. The fluid from the wound is collected into a container. The benefits of negative pressure wound therapy have been reported to include removal of infectious material, reduction in oedema and improved perfusion to tissue. Since few years, a new negative pressure wound therapy has been created for closed wounds to reduce time of healing and avoid wound complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* ≥10cm emergency median laparotomy
* Abdominal wall and skin closure in first intent
* Septic peritoneal cavity (purulent and/or fecaloid free liquid and/or abscess)
* Informed written consent

Exclusion Criteria:

* No abdominal wound closure in first intent
* Allergy or hypersensitivity to silver
* Application of a mesh for abdominal wall closure
* Patients under corticosteroids or other immunosuppressive treatment.
* Women who are pregnant or breast-feeding.
* Intention to become pregnant during the course of the study.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Previous enrolment in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
To determine if the use of prophylactic negative-pressure wound therapy (Prevena) reduces the incidence of superficial surgical site infection after emergency laparotomy in patients at high-risk for SSI | up to 30 days post procedure
  Any SSI may cause redness, delayed healing, fever, pain, tenderness, warmth, or swelling. Superficial site infection will be assessed by Wound Classification System Using the American College of Surgeons National Surgical Quality Improvement Program ACS-NSQIP :
  * Clean; these are uninfected operative wounds in which no inflammation.
  * Clean/contaminated; These are operative wounds in which the respiratory, alimentary, genital, or urinary tract is entered Under controlled conditions and without unusual contamination.
  * Contaminated; These include open, fresh, accidental wounds, operations with major breaks in sterile technique or gross spillage from the gastrointestinal tract, and incisions in which acute, non-purulent inflammation is encountered.
  * Dirty ; These include old traumatic wounds with retained devitalized tissue and those that involve existing clinical infection or perforated viscera.

SECONDARY OUTCOMES:
Length of stay (LOS) in days. | 30 days post procedure
  LOS is defined as days from operation to discharge; 30d LOS is defined as the index LOS plus all readmission days within 30d related to any wound complications.
30-day Return to Operating Room (ROR) | 30 days post procedure
  Reoperation for wound complication within 30 days involving incision and drainage in the operating room; opening the skin to drain a superficial soft tissue infection at bedside or in the office is not considered reoperation.
Incidence rates of wound complications | 30 days post procedure
  Individual rates of the incidence of each of the following: dehiscence (skin or fascia), seroma, lymph leak, infection, hematoma, ischemia and necrosis.

OTHER OUTCOMES:
A rate of parietal incisional hernia apparition after surgery | 2 years post procedure
  This complication rate is multifactorial can be related to:
  * An wall abcess
  * Obesity with a BMI > 35 Kg/m2
  * medications
  * Malnutrition
  * Being an elderly adult
  * Smoking
  * Cancer
  * a weak immune system
  * diabetes

REFERENCES:
- [Result] Conde-Green A, Chung TL, Holton LH 3rd, Hui-Chou HG, Zhu Y, Wang H, Zahiri H, Singh DP. Incisional negative-pressure wound therapy versus conventional dressings following abdominal wall reconstruction: a comparative study. Ann Plast Surg. 2013 Oct;71(4):394-7. doi: 10.1097/SAP.0b013e31824c9073. PMID 22868327
- [Result] Gorgulu T. A Complication of Management of Closed Incision with Negative-Pressure Wound Therapy. Aesthet Surg J. 2015 Jul;35(5):NP113-5. doi: 10.1093/asj/sju120. Epub 2015 May 29. No abstract available. PMID 26026135
- [Result] Dohmen PM, Misfeld M, Borger MA, Mohr FW. Closed incision management with negative pressure wound therapy. Expert Rev Med Devices. 2014 Jul;11(4):395-402. doi: 10.1586/17434440.2014.911081. Epub 2014 Apr 22. PMID 24754343
- [Result] Ingargiola MJ, Daniali LN, Lee ES. Does the application of incisional negative pressure therapy to high-risk wounds prevent surgical site complications? A systematic review. Eplasty. 2013 Sep 20;13:e49. eCollection 2013. PMID 24106562
- [Result] Wilkes RP, Kilpad DV, Zhao Y, Kazala R, McNulty A. Closed incision management with negative pressure wound therapy (CIM): biomechanics. Surg Innov. 2012 Mar;19(1):67-75. doi: 10.1177/1553350611414920. Epub 2011 Aug 25. PMID 21868417
- [Result] Vargo D. Negative pressure wound therapy in the prevention of wound infection in high risk abdominal wound closures. Am J Surg. 2012 Dec;204(6):1021-3; discussion 1023-4. doi: 10.1016/j.amjsurg.2012.10.004. PMID 23231938
- [Result] Zaidi A, El-Masry S. Closed-incision negative-pressure therapy in high-risk general surgery patients following laparotomy: a retrospective study. Colorectal Dis. 2017 Mar;19(3):283-287. doi: 10.1111/codi.13458. PMID 27416813
- [Result] Gunatilake RP, Swamy GK, Brancazio LR, Smrtka MP, Thompson JL, Gilner JB, Gray BA, Heine RP. Closed-Incision Negative-Pressure Therapy in Obese Patients Undergoing Cesarean Delivery: A Randomized Controlled Trial. AJP Rep. 2017 Jul;7(3):e151-e157. doi: 10.1055/s-0037-1603956. Epub 2017 Jul 14. PMID 28717587
- [Result] Reddix RN Jr, Tyler HK, Kulp B, Webb LX. Incisional vacuum-assisted wound closure in morbidly obese patients undergoing acetabular fracture surgery. Am J Orthop (Belle Mead NJ). 2009 Sep;38(9):446-9. PMID 19911098
- [Result] Stannard JP, Volgas DA, McGwin G 3rd, Stewart RL, Obremskey W, Moore T, Anglen JO. Incisional negative pressure wound therapy after high-risk lower extremity fractures. J Orthop Trauma. 2012 Jan;26(1):37-42. doi: 10.1097/BOT.0b013e318216b1e5. PMID 21804414
- [Result] Pauser J, Nordmeyer M, Biber R, Jantsch J, Kopschina C, Bail HJ, Brem MH. Incisional negative pressure wound therapy after hemiarthroplasty for femoral neck fractures - reduction of wound complications. Int Wound J. 2016 Oct;13(5):663-7. doi: 10.1111/iwj.12344. Epub 2014 Aug 14. PMID 25125244
- [Result] Redfern RE, Cameron-Ruetz C, O'Drobinak SK, Chen JT, Beer KJ. Closed Incision Negative Pressure Therapy Effects on Postoperative Infection and Surgical Site Complication After Total Hip and Knee Arthroplasty. J Arthroplasty. 2017 Nov;32(11):3333-3339. doi: 10.1016/j.arth.2017.06.019. Epub 2017 Jun 17. PMID 28705547
- [Result] Hansen E, Durinka JB, Costanzo JA, Austin MS, Deirmengian GK. Negative pressure wound therapy is associated with resolution of incisional drainage in most wounds after hip arthroplasty. Clin Orthop Relat Res. 2013 Oct;471(10):3230-6. doi: 10.1007/s11999-013-2937-3. PMID 23539123
- [Result] Semsarzadeh NN, Tadisina KK, Maddox J, Chopra K, Singh DP. Closed Incision Negative-Pressure Therapy Is Associated with Decreased Surgical-Site Infections: A Meta-Analysis. Plast Reconstr Surg. 2015 Sep;136(3):592-602. doi: 10.1097/PRS.0000000000001519. PMID 26313829
- [Result] Wiegering A, Dietz UA, Corteville C, Plassmeier L, Jurowich C, Germer CT, Krajinovic K. Impact of incisional negative pressure wound therapy on perineal wound healing after abdominoperineal rectum extirpation. Int J Colorectal Dis. 2017 Feb;32(2):291-293. doi: 10.1007/s00384-016-2704-5. Epub 2016 Nov 14. PMID 27844201
- [Result] Bonds AM, Novick TK, Dietert JB, Araghizadeh FY, Olson CH. Incisional negative pressure wound therapy significantly reduces surgical site infection in open colorectal surgery. Dis Colon Rectum. 2013 Dec;56(12):1403-8. doi: 10.1097/DCR.0b013e3182a39959. PMID 24201395
- [Result] Webster J, Liu Z, Norman G, Dumville JC, Chiverton L, Scuffham P, Stankiewicz M, Chaboyer WP. Negative pressure wound therapy for surgical wounds healing by primary closure. Cochrane Database Syst Rev. 2019 Mar 26;3(3):CD009261. doi: 10.1002/14651858.CD009261.pub4. PMID 30912582
- [Result] Zwanenburg PR, Tol BT, Obdeijn MC, Lapid O, Gans SL, Boermeester MA. Meta-analysis, Meta-regression, and GRADE Assessment of Randomized and Nonrandomized Studies of Incisional Negative Pressure Wound Therapy Versus Control Dressings for the Prevention of Postoperative Wound Complications. Ann Surg. 2020 Jul;272(1):81-91. doi: 10.1097/SLA.0000000000003644. PMID 31592899
- [Result] Moher D, Shamseer L, Clarke M, Ghersi D, Liberati A, Petticrew M, Shekelle P, Stewart LA; PRISMA-P Group. Preferred reporting items for systematic review and meta-analysis protocols (PRISMA-P) 2015 statement. Syst Rev. 2015 Jan 1;4(1):1. doi: 10.1186/2046-4053-4-1. PMID 25554246